CLINICAL TRIAL: NCT03004651
Title: Impact of Body Mass Index on the Agreement Between Ultrasound- and Clinical Assessments of Disease Activity in RA : Cross-sectionnal Study
Brief Title: BMI and Ultrasound/Clinical Assessments of RA Disease Activity
Acronym: RABODI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Pitié-Salpêtrière Hospital (Other); Hospital Ambroise Paré Paris (Other); Nantes University Hospital (Other); Rennes University Hospital (Other); University Hospital, Grenoble (Other); CHU Brest Hôpital La Cavale Blanche (Unknown); Hospital Purpan (Other); Centre Hospitalier Lyon Sud (Other); Central Hospital, Nancy, France (Other); Centre Hospitalier de la côte Basque (Other)
Responsible Party: Sponsor
Other Study IDs: 9742
Record Dates: First submitted 2016-12-07; First posted 2016-12-29 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Obsessional Erotomania

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese Patients: Power Doppler ultrasound on obese patients with PR comparating with a clinical evaluation (swollen joint count (SJC) as componant of SDAI)
  Interventions: Other: Power Doppler ultrasound; Other: Clinical evaluation
- Non obese patients: Power Doppler ultrasound on non obese patients with PR comparating with a clinical evaluation (swollen joint count (SJC) as componant of SDAI)
  Interventions: Other: Power Doppler ultrasound; Other: Clinical evaluation

INTERVENTIONS:
Other: Power Doppler ultrasound — Mesure of synovitis (≥ grade 1 synovitis on a semi-quantitative scale)
Other: Clinical evaluation — swollen joint count (SJC) as componant of SDAI

SUMMARY:
Comparison of the level of agreement between Power Doppler ultrasound measured number of synovitis (≥ grade 1 on a semi-quantitative scale) and clinically defined number of swollen joints in obese (i.e. BMI>30) versus normally weighted RA patients.

DETAILED DESCRIPTION:
Clinical evaluation of synovitis in rheumatoid arthritis (RA) is difficult in obese and overweighted patients, due to the fat pad located around the joint, that can over- or under estimate the number of joints regarded as swollen by clinical examination. RA in obese and overweighted patients has several distinctive characteristics as compared to the disease observed in normally weighted subjects: diease activity (assessed by composites scores such as Disease Activity Score (DAS28) or Simple Disease Activity Index (SDAI)) is higher, while response to treatment and severity (asessed by radiographic progression) are lower.

Objectives:

Primary end point: Comparison of the level of agreement between the number of joints considered abnormal by Power Doppler ultrasound synovitis (≥ grade 1 on a semi-quantitative scale) and clinical examination (swollen joint count (SJC) as componant of SDAI) in obese (i.e. BMI>30) versus normally weighted RA patients.

Secondary end points :

* Comparison of the level of agreement between clinical and ultrasound findings in overweighted versus normally weighted patients, when joint count evaluation is based on another composite index ((DAS28-CRP et DAS44-CRP), based on the number of tender joints, and based on a joint by joint evaluation
* Comparison of agreement between obese and non obese
* Evaluation of the impact of other factors than BMI on the level of agreement between Power Doppler ultrasound defined number of synovitis and clinically defined swollen joint count
* Reliability between Ultrasound and clinical examination across the different investigation centers Study design: prospective multicenter observational study Inclusion criteria: RA patients fulfilling ACR/EULAR 2010 criteria Exclusion criteria: patient simultaneously included in another study with blinded treatment; Steinbrocker class IV patients Outcome measure : Level of agreement between SJC and power Doppler US synovitis

ELIGIBILITY:
Inclusion criteria:

* RA patients fulfilling ACR/EULAR 2010 criteria

Exclusion criteria:

* Patient simultaneously included in another study with blinded treatment; Steinbrocker class IV patients, pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical evaluation of synovitis in rheumatoid arthritis (RA) is difficult in obese and overweighted patients, due to the fat pad located around the joint, that can over- or under estimate the number of joints regarded as swollen by clinical examination.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Comparison of the level of agreement between the number of abnormal joints and clinical evaluation | 18 months
  Comparison of the level of agreement between the number of abnormal joints as defined by Power Doppler ultrasound (≥ grade 1 synovitis on a semi-quantitative scale) and clinical evaluation (swollen joint count (SJC) as componant of SDAI) in obese

SECONDARY OUTCOMES:
Comparison of the level of agreement between clinical and ultrasound findings on function of patient's weight | 18 months
  Comparison of the level of agreement between clinical and ultrasound findings in overweighted versus normally weighted patients, when joint count evaluation is based on another composite index ((DAS28-CRP et DAS44-CRP), based on the number of tender joints, and based on a joint by joint evaluation
Impact of other factors on the level of agreement between Power Doppler ultrasound and clinical exam | 18 months
  Evaluation of the impact of other factors than BMI on the level of agreement between Power Doppler ultrasound defined number of synovitis and clinically defined swollen joint count
Reproducibility of the comparison between Ultrasound and clinical examination | 18 months
  Reliability between Ultrasound and clinical examination across the different investigation centers

CONTACTS AND LOCATIONS:
Overall Officials: Gaël MOUTERDE, PH, Principal Investigator — CHU de Montpellier
Locations (1):
- University Regional Hospital Lapeyronie, Montpellier, Languedoc-Roussillon, France

IPD SHARING:
Plan to Share IPD: No